CLINICAL TRIAL: NCT05089526
Title: Opioid-free Anesthesia With a Mixture of Dexmedetomidine-lidocaine-ketamine in Laparoscopic Cholecystectomies
Brief Title: Opioid-free Anesthesia in Laparoscopic Cholecystectomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: lap-chol-opioid free
Record Dates: First submitted 2021-10-10; First posted 2021-10-22 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chronic; Cholecystectomy; Ketamine; Dexmedetomidine; Lidocaine; Central Nervous System Depressants; Analgesia; Analgesics; Analgesic Non-narcotic
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Agnosia | interventions — Fentanyl; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine-lidocaine-dexmedetomidine (KLD) group (Active Comparator): combination of ketamine-lidocaine-dexmedetomidine in one syringe
  Interventions: Drug: ketamine-lidocaine-dexmedetomidine
- fentanyl (control) group (Active Comparator): syringe of fentanyl
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: ketamine-lidocaine-dexmedetomidine — In the KLD group, patients will be administered 0,25 mcg/kg Dexmedetomidine in 100 mL of normal saline within 10 minutes. Followingly, they will receive 1mL/10 kg of the solution containing ketamine, lidocaine and dexmedetomidine at predefined concentrations. As maintenance, they will be receiving
  1mL/10kg/h of the aforementioned solution.
  Other Names: KLD group
  Arms: ketamine-lidocaine-dexmedetomidine (KLD) group
Drug: fentanyl — In the fentanyl group, patients will be administered 2 mcg/kg fentanyl in 100 mL of normal saline within 10 minutes. Followingly, they will receive 1mL/10 kg of normal saline solution 0.9%. As maintenance, they will be receiving 1mL/10kg/h of normal saline solution 0.9%.
  Other Names: Control group
  Arms: fentanyl (control) group

SUMMARY:
The aim of this study will be to investigate the effect of an opioid-free anesthesia regimen with a mixture of dexmedetomidine-lidocaine-ketamine in the same syringe versus fentanyl analgesia in elective laparoscopic cholecystectomies

DETAILED DESCRIPTION:
Inadequately treated postoperative pain after laparoscopic cholecystectomy may untowardly affect early recovery and also lead to the development of chronic pain. Laparoscopic surgery is associated with diminished postoperative pain but this does not mean that patients subjected to laparoscopic operations are not in need for analgesia intra- and postoperatively. Pneumoperitoneum can lead to postoperative discomfort and occasionally intense postoperative shoulder pain. Opioid-based analgesia is associated with side-effects, such as respiratory depression, postoperative nausea and vomiting and occasional induction of tolerance and hyperalgesia.

Therefore, in recent years research has focused on the quest for non-opioid-based regimens for perioperative analgesia in the context of multimodal analgesic techniques. These techniques have been shown to possess significant advantages, such as allowing earlier mobilization after surgery, early resumption of enteral feeding and reduced hospital length of stay. In this context, the intraoperative intravenous injection of lidocaine has been reported to improve postoperative pain control, reduce opioid consumption and improve the quality of postoperative functional recovery after general anesthesia. Intraoperative infusions of ketamine (an N-methyl-D-aspartate receptor inhibitor) have also been correlated with reduced pain scores and a decrease in analgesic requirements postoperatively. Lastly, dexmedetomidine is a highly selective alfa-2 adreno-ceptor agonist that provides sedation, analgesia, and sympatholysis. Its perioperative intravenous administration has been associated with a reduction in postoperative pain intensity, analgesic consumption and nausea. There is insufficient data in literature investigating the effect of combinations of these agents intraoperatively. It would be of interest to demonstrate whether the administration of combinations can be used towards the achievement of a completely opioid-free anesthetic regimen. Additionally, it can be hypothesized that the combination of non-opioid drugs with different targets can lead to enhanced postoperative recovery, an improved opioid-sparing effect and a decrease in the development of chronic pain as compared to the administration of opioids. Therefore, the aim of this study will be to investigate the effect of a combination of intravenous infusions of lidocaine-ketamine-dexmedetomidine versus fentanyl on recovery profile and postoperative pain after elective laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* American Society of Anesthesiologists (ASA) classification I-II
* elective laparoscopic cholecystectomy

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2
* contraindications to local anesthetic administration or non-steroidal agents administration
* systematic use of analgesic agents preoperatively
* chronic pain syndromes preoperatively
* neurological or psychiatric disease on treatment
* pregnancy
* severe hepatic or renal disease
* history of cardiovascular diseases/ arrhythmias/ conduction abnormalities
* bradycardia(<55 beats/minute)
* drug or alcohol abuse
* language or communication barriers lack of informed consent

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score at discharge from Post-Anesthesia Care Unit (PACU) | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  pain score by the use of Numeric Rating Scale (NRS) at discharge from PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 3 hours postoperatively | 3 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 3 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

SECONDARY OUTCOMES:
Post Anesthesia Care Unit (PACU) duration of stay | immediately postoperatively
  duration of patient stay at PACU
sedation on arrival to Post-Anesthesia Care Unit | immediately postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
sedation at discharge from Post-Anesthesia Care (PACU) Unit | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
sevoflurane consumption during general anesthesia | change of sevoflurane vaporizer weight from before induction to end of anesthesia, an average period of 1-2 hours
  the sevoflurane vaporizer will be weighed before anesthetic induction and at the end of anesthesia and consequently sevoflurane consumption during anesthesia will be determined
time to first request for analgesia | during stay in Post-Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  the time for the first patient request for analgesia will be noted
morphine consumption in Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  mg of morphine requested during patient PACU stay
tramadol consumption in the first 24 hours | 24 hours postoperatively
  patients will be followed for cumulative tramadol consumption for 24 hours postoperatively
sleep quality | 24 hours postoperatively
  subjective evaluation of sleep quality by patients, based on a sleep questionnaire (evaluation of sleep duration, number of nocturnal awakenings and marking of sleep quality
first mobilization after surgery | 24 hours postoperatively
  patients will be questioned regarding the time at which they mobilized after surgery
gastrointestinal recovery after surgery | 24 hours postoperatively
  patients will be questioned regarding the time they first felt enteral sounds and the time they had their first flatus after surgery
satisfaction from postoperative analgesia | 24 hours postoperatively
  satisfaction from postoperative analgesia on a six-point Likert scale with 1 marked as minimal satisfaction and 6 as maximal satisfaction
first fluid intake | 24 hours postoperatively
  patients will be questioned regarding the time they had their first fluid intake
first solid intake | 24 hours postoperatively
  patients will be questioned regarding the time they had their first solid intake
hospitalization time | 96 hours postoperatively
  duration of hospital stay after surgery in hours
fentanyl requirement during surgery | intraoperatively
  dose of required fentanyl intraoperatively to maintain systolic arterial blood pressure and heart rate within the 20% of baseline value
side effects intraoperatively | intraoperatively
  patients will be monitored for side-effects of the administered agents intraoperatively
side effects postoperatively | 48 hours postoperatively
  patients will be monitored for side-effects of the administered agents postoperatively
incidence of chronic pain 1 month after surgery | 1 month after surgery
  occurrence of chronic pain at the site of the operation 1 month after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement
incidence of chronic pain 3 months after surgery | 3 months after surgery
  occurrence of chronic pain at the site of the operation 3 months after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement

OTHER OUTCOMES:
time to emergence | up to 2-3 hours after start of surgery
  time from sevoflurane discontinuation to first patient response (eye opening)
time to extubation | up to 2-3 hours after start of surgery
  time from sevoflurane discontinuation to tracheal extubation

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Evangelismos General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavand'homme P, Steyaert A. Opioid-free anesthesia opioid side effects: Tolerance and hyperalgesia. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):487-498. doi: 10.1016/j.bpa.2017.05.003. Epub 2017 May 17. PMID 29739537
- [Background] Frauenknecht J, Kirkham KR, Jacot-Guillarmod A, Albrecht E. Analgesic impact of intra-operative opioids vs. opioid-free anaesthesia: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):651-662. doi: 10.1111/anae.14582. Epub 2019 Feb 25. PMID 30802933
- [Background] Lavand'homme P, Estebe JP. Opioid-free anesthesia: a different regard to anesthesia practice. Curr Opin Anaesthesiol. 2018 Oct;31(5):556-561. doi: 10.1097/ACO.0000000000000632. PMID 29994942
- [Background] Mulier J. Opioid free general anesthesia: A paradigm shift? Rev Esp Anestesiol Reanim. 2017 Oct;64(8):427-430. doi: 10.1016/j.redar.2017.03.004. Epub 2017 Apr 18. No abstract available. English, Spanish. PMID 28431750
- [Background] Mauermann E, Ruppen W, Bandschapp O. Different protocols used today to achieve total opioid-free general anesthesia without locoregional blocks. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):533-545. doi: 10.1016/j.bpa.2017.11.003. Epub 2017 Nov 24. PMID 29739542
- [Background] Panchgar V, Shetti AN, Sunitha HB, Dhulkhed VK, Nadkarni AV. The Effectiveness of Intravenous Dexmedetomidine on Perioperative Hemodynamics, Analgesic Requirement, and Side Effects Profile in Patients Undergoing Laparoscopic Surgery Under General Anesthesia. Anesth Essays Res. 2017 Jan-Mar;11(1):72-77. doi: 10.4103/0259-1162.200232. PMID 28298760
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Toleska M, Dimitrovski A. Is Opioid-Free General Anesthesia More Superior for Postoperative Pain Versus Opioid General Anesthesia in Laparoscopic Cholecystectomy? Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2019 Oct 1;40(2):81-87. doi: 10.2478/prilozi-2019-0018. PMID 31605587
- [Background] Saadawy IM, Kaki AM, Abd El Latif AA, Abd-Elmaksoud AM, Tolba OM. Lidocaine vs. magnesium: effect on analgesia after a laparoscopic cholecystectomy. Acta Anaesthesiol Scand. 2010 May;54(5):549-56. doi: 10.1111/j.1399-6576.2009.02165.x. Epub 2009 Nov 16. PMID 19919581
- [Background] Lu J, Wang JF, Guo CL, Yin Q, Cheng W, Qian B. Intravenously injected lidocaine or magnesium improves the quality of early recovery after laparoscopic cholecystectomy: A randomised controlled trial. Eur J Anaesthesiol. 2021 Mar 1;38(Suppl 1):S1-S8. doi: 10.1097/EJA.0000000000001348. PMID 33074940
- [Background] Bakan M, Umutoglu T, Topuz U, Uysal H, Bayram M, Kadioglu H, Salihoglu Z. Opioid-free total intravenous anesthesia with propofol, dexmedetomidine and lidocaine infusions for laparoscopic cholecystectomy: a prospective, randomized, double-blinded study. Braz J Anesthesiol. 2015 May-Jun;65(3):191-9. doi: 10.1016/j.bjane.2014.05.001. Epub 2014 Jun 3. PMID 25925031